CLINICAL TRIAL: NCT02876250
Title: Postconditioning by Cyclosporin A in Pulmonary Transplantation
Acronym: CsA Poumon
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-816
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Lung Transplantation
Keywords: Lung transplantation; Cyclosporine; Postconditioning
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cyclosporine A (Experimental): a pharmacological postconditioned group with IV administration of 2.5 mg/kg of CsA prior to first graft reperfusion
  Interventions: Drug: Cyclosporine A
- Control (Placebo Comparator): a control group with IV administration of 2.5 mg/kg of placebo prior to first graft reperfusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine A — a pharmacological postconditioned group with IV administration of 2.5 mg/kg of CsA prior to first graft reperfusion
  Arms: Cyclosporine A
Drug: Placebo — a control group with IV administration of 2.5 mg/kg of placebo prior to first graft reperfusion
  Arms: Control

SUMMARY:
The morbidity and mortality of patients undergoing lung transplantation in the acute phase following surgical intervention is mainly due to the primary graft failure (PGF).

The occurrence of PGF is multi factorial but is mainly caused by ischemia-reperfusion injury. The pulmonary graft suffers two periods of ischemia one when it is explanted from the donor (cold ischemia) followed by another when it is grafted into the recipient's thoracic cavity (warm ischemia). The brutal reperfusion of the graft exposes it to reperfusion injury that causes PGF. PGF occurs in up to 20% of transplanted patients and is associated with significantly higher levels of 30-days all-cause mortality. Patients with PGF have a 40% mortality at 30-days versus a 6% mortality in patients without PGF.

Ischemic postconditioning, has recently been described in experimental models of ischemia-reperfusion injury in the heart, and although not yet fully understood. Several studies suggest that the mitochondria play a central role in cellular survival mechanisms after a prolonged period of ischemia-reperfusion (with the mitochondrial permeability transition pore (mPTP)).

Experimental studies have shown that cyclosporin A (CsA) administered prior to reperfusion binds to cyclophilin D and blocks the opening of mPTP after reperfusion. This protective effect of ischemia-reperfusion injury by CsA has been shown in experimental studies and in clinical phase II trials in reperfused myocardial infarction patients.

The hypothesis of this study is that the administration of CsA in transplanted patients (before re-opening of the first pulmonary graft vessels) protects the transplanted lung(s) from the deleterious effects of ischemia-reperfusion injury and thus reduce the frequency and severity of PGF.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old, man or woman, who are listed for pulmonary transplantation either mono or double lung transplantation.

Exclusion Criteria:

* No contra-indication to CsA administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio (ratio of arterial oxygen partial pressure to fractional inspired oxygen) | 2 hours post-lung transplantation
PaO2/FiO2 ratio | 6 hours post-lung transplantation
PaO2/FiO2 ratio | 12 hours post-lung transplantation
PaO2/FiO2 ratio | 18 hours post-lung transplantation
PaO2/FiO2 ratio | 24 hours post-lung transplantation
PaO2/FiO2 ratio | 36 hours post-lung transplantation
PaO2/FiO2 ratio | 48 hours post-lung transplantation
PaO2/FiO2 ratio | 60 hours post-lung transplantation
PaO2/FiO2 ratio | 72 hours post-lung transplantation

SECONDARY OUTCOMES:
primary graft failure grade | 72 hours
  clinical status of primary graft failure at 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: François TRONC, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No